CLINICAL TRIAL: NCT02563665
Title: A Prospective Study on Safety and Efficacy of Sofosbuvir Based Antiviral Regimen for Treating Hepatitis C in Patients With Moderate to Advanced Chronic Kidney Disease and Patients Receiving Renal Replacement Therapy
Brief Title: Safety and Efficacy of Sofosbuvir Based Antiviral Regimen for Treating Hepatitis C in Patients With Moderate to Advanced Chronic Kidney Disease and Patients Receiving Renal Replacement Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-HCKD/001/SOFO/2015
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2016-10

CONDITIONS: CKD With Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- advanced chronic kidney disease: Subjects on dialysis with GFR (Glomerular Filtration Rate) > 30
- Renal replacement therapy.: Subjects who are not on dialysis with GFR (Glomerular Filtration Rate) < 15

SUMMARY:
All patients with chronic kidney disease (stages 3, 4 and 5) and chronic dialysis patients with HCV infection attending nephrology and Hepatology OPD or getting outpatient dialysis at the dialysis unit of ILBS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe renal dysfunction (CKD stage 3, 4, 5) and chronic dialysis patients
2. Patients consented for the study protocol by signing the informed consent.

Exclusion Criteria:

1. Age less than 18 years
2. Confirmed pregnancy
3. HCV-HIV Co infection
4. HBV-HCV co infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic kidney disease (stages 3, 4 and 5) and chronic dialysis patients with Hepatitis C infection attending nephrology and Hepatology OPD (Out Patient Department) or getting outpatient dialysis at the dialysis unit of Institute of Liver and Biliary Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response 24 defined as HCV RNA <Lower Level of Qunatification 24 weeks after discontinuation of therapy. | 1 year

SECONDARY OUTCOMES:
number of adverse Events in both groups | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Suman Lata Nayak, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India